CLINICAL TRIAL: NCT05687682
Title: A Phase I, Open-Label, Dose-Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AM-928 Infusion in Subjects With Advanced Solid Tumors
Brief Title: Safety of AM-928 Infusion in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AcadeMab Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A928-CLN-001
Record Dates: First submitted 2023-01-07; First posted 2023-01-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor
Keywords: Solid tumor; EpCAM; Antibody

STUDY DESIGN:
Intervention Model Description: AM-928
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Level -1 (Experimental): 0.1 mg/kg
  Interventions: Biological: AM-928
- Level 1 (Experimental): 0.3 mg/kg (Starting Dose)
  Interventions: Biological: AM-928
- Level 2 (Experimental): 1 mg/kg
  Interventions: Biological: AM-928
- Level 3 (Experimental): 3 mg/kg
  Interventions: Biological: AM-928
- Level 4 (Experimental): 6 mg/kg
  Interventions: Biological: AM-928
- Level 5 (Experimental): 10 mg/kg
  Interventions: Biological: AM-928
- Level 6 (Experimental): 15 mg/kg
  Interventions: Biological: AM-928

INTERVENTIONS:
Biological: AM-928 — AM-928, which is a humanized anti-EpCAM monoclonal antibody developed by AcadeMab Biomedical Inc.

SUMMARY:
This is a Phase I, open-label, dose-escalation study for a novel cancer treatment, AM-928, intravenous infusion antibody for advanced solid tumor. The study is aimed to learn the safety, tolerability, pharmacokinetics, and preliminary efficacy profile of AM-928.

The dose escalation strategy will adopt accelerated titration combined with a Bayesian optimal interval (BOIN) design. Seven dose levels are designed and each participant will be assigned to a specific dose regimen depending on the time of enrollment. In the study, each participant will receive AM-928 treatment cycles till meeting any treatment discontinuation criterion and be followed for safety and long-term survival.

The whole study is expected to take approximately three years to complete.

DETAILED DESCRIPTION:
This is a first-in-human Phase I, open-label, dose-escalation study to investigate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of AM-928 infusion in subjects with advanced solid tumors in multiple sites in Taiwan.

Eligible subjects will be dosed with different dosages of AM-928 in 1 of the 7 dose levels (0.1, 0.3, 1, 3, 6, 10, 15 mg/kg). Dose levels will be escalated from dose Level 1 at 0.3 mg/kg to Level 6 at 15 mg/kg of AM-928 (or may be de-escalated to Level -1 at 0.1 mg/kg), which will be administered (intravenous infusion) once weekly (QW) for 4 weeks (D1, D8, D15, D22) as a treatment cycle until any treatment discontinuation criterion is met. Basically, there will be no breaks between dosing cycles. From Cycle 4, intra-subject dose escalation may be applied if supported by preliminary safety and PK data.

The dose escalation strategy will adopt accelerated titration combined with a Bayesian optimal interval (BOIN) design. The accelerated titration will be adopted for 0.3 mg/kg, while the BOIN design will be adopted for other dose levels, including 1 mg/kg, 3 mg/kg, 6 mg/kg, 10 mg/kg, and 15 mg/kg. In the "accelerated titration" stage, if any ≥ Grade 2 adverse event occurs, the current and subsequent dose groups will be changed to the BOIN dose escalation method. The target toxicity rate for the maximum tolerated dose (MTD) is ϕ= 0.3, and the maximum sample size is determined to be 30, maximum of 9 subjects per dose level. A cohort size of 3 and a maximum cohort number of 3 for each dose level will be adopted for subject recruitment. The dose escalation may end when one of the following criteria is met: (1) The planned sample size of 30 has been reached; (2) 9 subjects have been treated and evaluable for DLT at the next intended dose level (should not exceed 9 subjects at one dose level); (3) all doses explored appear to be overly toxic, and the MTD cannot be determined.

The Scientific Review Committee (SRC) will review the safety and/or efficacy data at the end of each dose level cohort for escalation or de-escalation decision (when the DLT rate indicates staying at the current dose, the review process may be waived). Besides, an emergency meeting will be held if the SRC has any safety concerns. A final review process is scheduled at the end of dose escalation for MTD determination. The dose with the toxicity rate closest to the target toxicity rate (ϕ= 0.3) will be selected as MTD.

If the SRC determines that the safety profile of a specific dose level is unfavorable for subjects, the SRC may eliminate that dose level even if the toxicity rate is below 0.3. In this case, the subsequent subjects will be enrolled into the lower dose level(s) following the BOIN design and the lower dose level with the toxicity rate closest to the target toxicity rate (ϕ= 0.3) will be selected as MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years
2. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors that are refractory to or intolerant of existing standard therapy, for which no effective standard therapy that confers clinical benefit is available
3. Availability of archival tissue specimens for EpCAM immunohistochemistry (IHC) staining. Tumor tissues acceptable include:

   - Tumor tissue sample collected at the time of initial diagnosis

   - The most recent available recurrent/metastatic tumor biopsy tissue if available (a pre-treatment biopsy is encouraged if the biopsy site is safely accessible) Note: this criterion is fulfilled if there is a qualified tumor sample (tumor cells were presented in the tumor biopsy tissue), and the tumor tissue slides can be obtained for IHC staining. It is not violated even if the staining result from biopsy obtained after the screening visit reveals that the slides contain no identifiable tumor cells.
4. Has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
6. Subject's life expectancy of at least 12 weeks
7. Has adequate hematopoietic, coagulation, hepatic function and renal function:

   - Hemoglobin ≥ 8.0 g/dL without transfusion or erythropoiesis stimulating agent support within 1 week
   * Absolute neutrophil count (ANC) ≥ 1,500 cells/μL without WBC growth factor support within 1 week
   * Total white blood cell (WBC) ≥ 2,500 cells/μL
   * Platelet ≥ 80,000 counts/μL without transfusion support within 1 week
   * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5× ULN and no sign of jaundice (≤ 3× ULN for subjects with known Gilbert disease)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3× ULN (≤ 5× ULN for subjects with tumor involvement in liver)
   * Serum albumin ≥ 3.0 g/dL
   * eGFR (CKD-EPI) ≥ 60 mL/min/1.73 m^2
8. A female subject with childbearing potential should be confirmed of not being pregnant or not lactating at the screening and during the study
9. Willingness and ability to comply with protocol-stated requirements, instructions, and restrictions in the investigator's judgement
10. Is able to understand the nature of this study and accepts to enter the study by signing written informed consent

Exclusion Criteria:

1. Received any localized cancer therapeutic modalities (e.g., surgery on target lesions, radiotherapy) within 4 weeks prior to initial dosing (except the palliative radiotherapy performed on non-target local lesions), or have any unrecovered surgical wound (except the wound from the biopsy at screening)
2. Received anti-tumor therapies such as chemotherapy, small molecular targeted therapy, hormone therapy, biological product therapy (mAbs, bispecific antibody, and ADC), or other anti-cancer agents within 2 weeks or 5 half-lives (whichever is shorter) before the first AM-928 dosing; received immunotherapy within 4 weeks or 5 half-lives (whichever is shorter) before the first AM-928 dosing.
3. Carries history of primary malignancy other than the entry diagnosis that could affect compliance with the protocol or interpretation of results within 3 years prior to the Screening Visit, except curatively treated non-melanoma skin cancer, cervical carcinoma in situ, or superficial bladder tumors
4. Received immunosuppressive medication(s) (including, but not limited to, steroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, tumor necrosis factor-ɑ antagonists, and calcineurin inhibitors) within 2 weeks (for those half-life ≤ 72 hours) or 4 weeks (for those half-life > 72 hours) prior to study dosing and during the study period, with the following caveats:

   - For steroids, ≤10 mg of prednisone per day or equivalent is allowed
   * Topical, ocular, intra-articular, intranasal, and inhaled corticosteroids is allowed. For a subject under long-term treatment of a concurrent disease/status, the dose should be stable (i.e., no change or decreasing dose) within 3 months prior to C1D1
   * The use of inhaled corticosteroids is allowed if they are on a stable dose (i.e., no change or decreasing dose within 3 months prior to C1D1)
   * The use of oral mineralocorticoids is allowed
   * Physiologic doses of corticosteroids for adrenal insufficiency or supportive care for a subject's advanced tumor may be allowed at the investigator's discretion
5. Subject with significant cardiopulmonary abnormalities as defined by:

   * Poorly controlled hypertension (systolic blood pressure > 150 mm-Hg and/or diastolic blood pressure > 100 mm-Hg on anti-hypersensitive medications)
   * Left ventricular ejection fraction (LVEF) < 50% at screening
   * History of symptomatic congestive heart failure > class 2 per New York Heart Association (NYHA) classification
   * History of myocarditis
   * Myocardial ischemia/infarction or unstable angina within 6 months of study enrollment
   * Uncontrolled serious cardiac arrhythmias
   * Corrected QT interval > 470 ms demonstrated by at least 2 ECGs > 30 minutes apart
   * Evidence of active pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or history of idiopathic pulmonary fibrosis. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
   * History of 2nd or 3rd-degree atrioventricular conduction defects
6. History of thromboembolic or cerebrovascular events within the last 6 months at screening, including transient ischemic attack, cerebrovascular accident, or deep vein thrombosis
7. Prior treatment with any EpCAM-targeted anti-cancer therapies
8. Subjects with the following infections:

   - History of active pulmonary tuberculosis infection ≤ 48 weeks prior to C1D1, regardless of treatment
   * Any major episode of infection requiring treatment with systemic antibiotics or hospitalization within 2 weeks prior to C1D1
   * Known human immunodeficiency virus (HIV) history
   * Presence of hepatitis B surface antigen (HBsAg) with HBV viral load > 2000 IU/mL (HBsAg-positive subjects with HBV viral load ≤ 2000 IU/mL are eligible. These subjects should continue to receive antiviral treatment during the study treatment and follow local HBV antiviral treatment standards after the study treatment during the study)
   * HCV RNA positive (subjects with a history of HCV infection are eligible if their HCV viral load cannot be detected at screening; curative antiviral therapy should have been completed at least 4 weeks before C1D1)
9. Administration of a live, attenuated vaccine within 4 weeks before C1D1 or anticipation that such a live, attenuated vaccine will be required during the study
10. Received any investigational product within 4 weeks before C1D1
11. History of severe allergic, anaphylactic, or other hypersensitivity reactions to humanized antibodies
12. Known hypersensitivity to any of the components of AM-928
13. Has unstable/uncontrolled central nervous system (CNS) malignancy, leptomeningeal, or brain metastasis (progressing or those who continue to require glucocorticoids or intrathecal chemotherapy)
14. Has symptomatic pleural effusion, pericardial effusion, or poorly controlled ascites
15. Suffering from side/toxic effects of previous or current therapy [i.e., National Cancer Institute - Common Terminology Criteria for Adverse Event (NCI-CTCAE) ≥ Grade 2] that, judged by the investigator, may interfere with the trial results or the subject's safety
16. Prior allogeneic stem cell, solid organ, or bone marrow transplantation
17. Subject with any underlying medical, mental, or psychological conditions that would impair the treatment compliance, contraindicate the use of the investigational product, or that may render the subject at high risk from treatment complications, in the opinion of the investigator, would not permit to participate in the study
18. All male subjects and female subjects with childbearing potential (between puberty and 1 year after menopause) should use at least one of the appropriate contraception methods shown below from signing ICF to at least 4 months or 5 half-lives (if data available), whichever is longer, after stopping study treatment.

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
    4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

    d.1. Use oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example, hormone vaginal ring or transdermal hormone contraception.

    d.2. Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) | Up to 29 days
  The MTD is defined the highest dose level that is closely to the toxicity rated defined in the study.
The incidence of dose-limiting toxicity (DLT) | Up to 29 days
  The DLT is specified treatment-emergent events that occur in cycle 1 treatment period, graded by NCI-CTCAE v5.0, and causality to study drug cannot be clearly ruled out.

SECONDARY OUTCOMES:
Number of participants with abnormalities in Laboratory Values | Up to 28 days after the last dose
  Number of participants with abnormal hematology (RBC, WBC with differentials (neutrophils, lymphocytes, monocytes, eosinophils, and basophils), platelet count, hemoglobin, and hematocrit), biochemistry (Albumin, total cholesterol, total bilirubin, direct bilirubin, alkaline phosphatase (ALP), AST, ALT, gamma-glutamyl transferase (γ-GT), total protein, blood urea nitrogen (BUN), lactate dehydrogenase (LDH), creatine kinase (CK), creatinine, estimated glomerular filtration rate (eGFR; 2021 CKD-EPI), triglyceride, amylase, lipase, glucose, uric acid, bicarbonate, calcium, chloride, inorganic phosphorus, iron, magnesium, potassium, and sodium), coagulation (prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR)), urinalysis (specific gravity, pH, occult blood, leukocytes, glucose, protein, ketones, bilirubin, and urine sediment (RBC, WBC, casts, epithelial cells, crystal, and microorganism)), and Troponin-T results
Number of treatment-emergent adverse events (TEAEs) | Up to 28 days after the last dose
  The TEAE is defined as adverse event (AE) occurred after the study drug administration. All TEAE will be assessed for severity by the investigator based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Incidence of subjects experiencing treatment-related AE with ≥ Grade 3 | Up to 28 days after the last dose
  The TEAE is defined as adverse event (AE) occurred after the study drug administration. All TEAE will be assessed for severity by the investigator based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Incidence of subjects experiencing infusion-related reaction | Day 1, Day 8, Day 15, Day 22 of Cycle 1 treatment
  The infusion-related reaction is adverse reaction due to study drug and occurred during an infusion and for 2 hours after the infusion completes. The symptom includes but not limited to fever, hypotension, hypertension, rash, nausea, dizziness.
Incidence of all-grade and Grade 3-4 laboratory abnormalities | Up to 28 days after the last dose
  The grading of the laboratory abnormalities is assessed based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Percentage of subjects tolerated at least 75% of the intended dose per cycle | Up to 3 months
  A subject will be treated weakly, 4 doses in a cycle
Number of participants with physical abnormalities | Up to 3 months
  Physical examination includes the following items: general appearance, skin, eyes, ears, nose, throat, head and neck (including thyroid), heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological system, and other body systems if applicable for describing the status of the subject's health.
Number of participants with chest x-ray abnormalities | Up to 3 months
  The chest x-ray will be evaluated by the investigators and noted as "normal", "NCS" or "CS".
Number of participants with abnormalities in vital signs | Up to 28 days after the last dose
  Vital signs measurement will consist of systolic/diastolic blood pressure, respiratory rate, pulse rate, body temperature, and oxygen saturation (SpO2).
Number of participants with abnormalities in 12-lead electrocardiogram (ECG) for each post-treatment evaluation until the end of Cycle 3 | Up to 3 months
  The results of ventricular rate, PR interval, QRS interval, QT interval, and QTc interval will be recorded.
AM-928 serum concentration | Day 1, 2, 3, 4, 8 and 15 of Cycle 1 treatment, Day 1 and 15 of Cycle 2, Day 1 of the following Cycle 3 and Cycle 5, and in 7 days after the last dose
  The serum concentration of AM-928
AM-928 Pharmacokinetic Parameter - Cmax | Week 1
  The peak post-dose concentration
AM-928 Pharmacokinetic Parameter - Tmax | Week 1
  Time at which Cmax is observed
AM-928 Pharmacokinetic Parameter - T 1/2 | Week 1
  Terminal phase elimination half-life
AM-928 Pharmacokinetic Parameter - AUC last | Week 1
  Area under the serum concentration-time profile (AUC) from time zero (T0) to the time of the last quantifiable concentration
AM-928 Pharmacokinetic Parameter - AUC 0-infinity | Week 1
  AUC from T0 extrapolated to infinite time
AM-928 Pharmacokinetic Parameter - CL | Week 1
  The volume of serum cleared of the drug per unit time.
AM-928 Pharmacokinetic Parameter - Vz | Week 1
  Volume of distribution
AM-928 Pharmacokinetic Parameter - Vss | Week 1
  Steady-state volume of distribution
AM-928 Pharmacokinetic Parameter - MRT | Week 1
  Mean Residence Time
AM-928 Pharmacokinetic Parameter - C trough | Day 8, Day 15, Day 22 of Cycle 1 treatment; Day 1, Day 15 of Cycle 2; Day 1 of Cycle 3 and Cycle 5
  The last pre-dose concentration at steady state before the next dose is administered
Objective response rate (ORR) | 6 months
  The proportion of treated subjects achieving the best overall response of Complete Response (CR) or Partial Response (PR) per RECIST 1.1
Disease control rate (DCR) | 6 months
  The proportion of treated subjects having achieved Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) per RECIST 1.1
Tumor growth rate (TGR) | Up to 28 days after the last dose
  The percent increase in the tumor volume per month
Tumor growth kinetics (TGK) | Up to 28 days after the last dose
  Change in the sum of the diameters of the target lesions per month
Change in Eastern Cooperative Oncology Group (ECOG) score | Up to 28 days after the last dose
  ECOG- Eastern Cooperative Oncology Group performance status is a scale used to assess how the disease affects the daily living abilities, and determine appropriate treatment and prognosis. It is a simple measure of functional status that determines ability of patient to tolerate therapies in cancer
Change in European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 score | Up to 28 days after the last dose
  The EORTC QLQ-C30 is a patient-reported outcome (PRO) questionnaire to assess the quality of life of cancer patients. Version 3.0 will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Pi-Chun Li, Ph.D., Study Director — AcadeMab Biomedical Inc.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No